CLINICAL TRIAL: NCT01359592
Title: A Phase II Trial of PET-Directed Therapy for Limited Stage Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: S1001 PET-Directed Therapy in Treating Patients With Limited-Stage Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000700624; S1001 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2011-05-21; First posted 2011-05-25 (Estimated); Results first posted 2021-06-30 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Lymphoma
Keywords: stage I adult diffuse large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; Fluorodeoxyglucose F18; Serotonin Plasma Membrane Transport Proteins; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PET Negative: R-CHOP (Active Comparator): R-CHOP x 3 Cycles
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Other: R-CHOP regimen; Other: laboratory biomarker analysis
- PET Positive: IFRT +Zevalin (Experimental): Standard IFRT+ Zevalin IV per ABW
  Interventions: Biological: rituximab; Other: laboratory biomarker analysis; Radiation: fludeoxyglucose F 18; Radiation: selective external radiation therapy; Radiation: yttrium Y 90 ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
  Arms: PET Negative: R-CHOP
Drug: doxorubicin hydrochloride
  Arms: PET Negative: R-CHOP
Drug: prednisone
  Arms: PET Negative: R-CHOP
Drug: vincristine sulfate
  Arms: PET Negative: R-CHOP
Other: R-CHOP regimen
  Arms: PET Negative: R-CHOP
Other: laboratory biomarker analysis
Radiation: fludeoxyglucose F 18
  Arms: PET Positive: IFRT +Zevalin
Radiation: selective external radiation therapy
  Arms: PET Positive: IFRT +Zevalin
Radiation: yttrium Y 90 ibritumomab tiuxetan
  Arms: PET Positive: IFRT +Zevalin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone, work in different ways to stop cancer cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill cancer cells. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Radiolabeled monoclonal antibodies, such as yttrium Y 90 ibritumomab tiuxetan, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Comparing results of diagnostic procedures, such as PET scan and CT scan, done before, during, and after chemotherapy may help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This phase II trial studies how well PET-directed chemotherapy works in treating patients with limited-stage diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the 5-year progression-free survival (PFS) rate in patients with newly diagnosed limited-stage diffuse, large B-cell lymphoma (DLBCL) using positron emission tomography (PET)/CT scan to direct therapy after 3 courses of rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone (R-CHOP).

Secondary

* To evaluate PFS within the PET-positive (+) and PET-negative (-) subgroups of patients with newly diagnosed limited-stage DLBCL.
* To evaluate toxicity of the protocol treatments in this patient population.
* To evaluate the response probability in this patient population.
* To evaluate overall survival in the overall population, and within the PET+ and PET- subgroups.
* To estimate the rate of upstaging at baseline by PET/CT at baseline among patients newly diagnosed with limited-stage DLBCL by CT imaging and to describe outcomes in patients upstaged by PET/CT at baseline to advanced DLBCL.
* To describe outcomes in the subgroup of patients upstaged by PET/CT.
* To evaluate the association of germinal center B-cell subtype (GCB) vs stromal-1 vs stromal-2 gene expression signatures with PFS or overall survival.

OUTLINE: This is a multicenter study. Patients are stratified according to whether the patient was upstaged to advanced stage DLBCL, based on local review of the baseline PET/CT (yes vs no).

Chemotherapy: Patients receive R-CHOP comprising rituximab IV, cyclophosphamide IV over 30-60 minutes, vincristine sulfate IV, and doxorubicin hydrochloride IV on day 1, and prednisone orally on days 1-5. Treatment repeats every 21 days for 3* courses. NOTE: *Patients found to have advanced stage DLBCL based on local review of the baseline PET scan receive 6 courses of R-CHOP.

FDG/PET - Radiotherapy: Patients undergo fludeoxyglucose F 18 positron emission tomography (FDG-PET)/CT scan at baseline, on days 15-18 of course 3, and at 12 weeks after completion of course 3. Patients with complete response (PET scan negative) receive one additional course of R-CHOP as above. Patients with partial response (PET scan positive) undergo involved-field radiotherapy (IFRT) 5 days a week for approximately 4-5 weeks.

Monoclonal antibody: Beginning 3-6 weeks after completion of IFRT, patients receive yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes and rituximab IV on day 1 and on day 7, 8, or 9.

Patients may undergo blood sample collection at baseline for correlative studies. Bone marrow tissue samples may be also collected for correlative studies.

After completion of study therapy, patients are followed up every 6 months for 2 years and then yearly for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients must have biopsy-proven diffuse large B-cell lymphoma (DLBCL)

  * Adequate sections or a paraffin block from the original diagnostic specimen must be submitted for review by the lymphoma pathology group
  * Lymphoma must express CD20 antigen by either flow cytometry using anti-CD20 antibodies or by immunoperoxidase staining of paraffin sections
  * Patients with primary mediastinal lymphoma or testicular lymphoma are not eligible
* Patients must have non-bulky stage I or II disease by Ann Arbor classification

  * This staging excludes FDG-PET evaluation
  * Patients who have stage I or II non-bulky disease on diagnostic CT scan, but are upstaged to stage III or IV based on FDG-PET evaluation, are also eligible
* Patients must have a diagnostic quality contrast-enhanced CT scan of the chest, abdomen, and pelvis AND baseline FDG-PET scan performed within 28 days prior to registration

  * Low-resolution "localization" CT scans performed as part of a combined PET/CT scan are not adequate for enrollment or response determination on this protocol
  * If a patient has an allergy to CT contrast, then a non-enhanced CT will be acceptable
* Patients must not have clinical evidence of central nervous system (CNS) involvement by lymphoma

  * Any laboratory or radiographic tests performed to assess CNS involvement must be negative and must be performed within 42 days prior to registration
* Patients may have either measurable or evaluable limited-stage DLBCL

  * Patients rendered free of measurable or evaluable disease by virtue of biopsy (resection) are also eligible
  * If patient has measurable disease it must be documented on the Lymphoma Baseline Tumor Assessment Form (Form #15187)
  * All measurable disease must be assessed within 28 days prior to registration
  * Patients with non-measurable disease in addition to measurable disease must have all non-measurable disease assessed within 42 days prior to registration
* Patients must have a unilateral or bilateral bone marrow biopsy performed within 42 days prior to registration

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 2 times upper limit of normal (ULN) (unless due to Gilbert syndrome)
* Patients must not be pregnant or nursing
* Women/men of reproductive potential must have agreed to use an effective contraceptive method during the study period
* Patients must not be known to be HIV-positive
* No other prior malignancy is allowed except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or II cancer from which the patient is currently in complete remission
  * Any other cancer from which the patient has been disease-free for 5 years

PRIOR CONCURRENT THERAPY:

* Patients must not have received prior chemotherapy, radiotherapy, or antibody therapy for lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2011-09; Primary Completion 2020-06-03 (Actual); Study Completion 2023-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O. Persky, MD, Principal Investigator — Yale University
Locations (240):
- United States (240):
  - Providence Cancer Center, Anchorage, Alaska
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Kaiser Permanente - Denver, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente - Lafayette, Lafayette, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Oncare Hawaii, Incorporated - Pali Momi, ‘Aiea, Hawaii
  - Leeward Radiation Oncology, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Parvin Radiation Oncology, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - MeritCare Broadway, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with nonbulky (< 10 cm) stage I/II untreated DLBCL received 3 cycles of standard R-CHOP therapy and underwent a centrally reviewed interim PET/computed tomography scan (iPET). Those with a negative iPET proceeded with 1 additional cycle of R-CHOP, whereas those with a positive iPET received involved field radiation therapy followed by ibritumomab tiuxetan radioimmunotherapy.
Groups:
- R-CHOP x 3: Chemotherapy for up to 3 cycles, 21 days/per cycle, with R-CHOP
  For each cycle, R-CHOP therapy included:
  Rituximab: 375 mg/m^2 IV administration on Day 1
  Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  Doxorubicin: 50 mg/m^2 IV administration on Day 1
  Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  Prednisone: 100 mg administered orally on Days 1 through 5
- R-CHOP x 6: Chemotherapy for up to 6 cycles, 21 days/per cycle, with R-CHOP
  For each cycle, R-CHOP therapy included:
  Rituximab: 375 mg/m^2 IV administration on Day 1
  Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  Doxorubicin: 50 mg/m^2 IV administration on Day 1
  Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  Prednisone: 100 mg administered orally on Days 1 through 5
- PET-negative: R-CHOP x 1: Chemotherapy for 1 cycle, 21 days/per cycle, with R-CHOP
  R-CHOP therapy included:
  Rituximab: 375 mg/m^2 IV administration on Day 1
  Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  Doxorubicin: 50 mg/m^2 IV administration on Day 1
  Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  Prednisone: 100 mg administered orally on Days 1 through 5
- PET-positive: IFRT + Yttrium-90 Ibritumomab Tiuxetan (Zevalin®): Patients start Involved-Field Radiation Therapy (IFRT) as soon as possible after the Day 15-18 PET/CT scan that follows Cycle 3 of R-CHOP, but no later than Day 35 after initiation of Cycle 3 of R-CHOP. Zevalin® treatment begins 3-6 weeks after Radiation Therapy is completed.
  Radiation Therapy included:
  IFRT: 180 cGy/day for a minimum dose of 3600 cGy and a maximum of dose of 4500 cGy
  Radioimmunotherapy included:
  Rituximab: 250 mg/m^2 IV administration on Day 1 then 7, 8, or 9
  Yttrium-90 ibritumomab tiuxetan: 0.4 mCi/kg or 0.3 mCi/kg, absolute maximum allowable dose of 32.0 mCi, 10 min IV infusion, on Day 7, 8 or 9
Period: Initial Registration
Arm/Group | R-CHOP x 3 | R-CHOP x 6 | PET-negative: R-CHOP x 1 | PET-positive: IFRT + Yttrium-90 Ibritumomab Tiuxetan (Zevalin®)
Started | 158 | 1 | 0 | 0
Eligible and Evaluable | 132 | 1 | 0 | 0
Completed | 129 | 1 | 0 | 0
Not Completed | 29 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Other reason not protocol specified | 1 | 0 | 0 | 0
Not completed — Ineligible | 26 | 0 | 0 | 0
Period: PET-Directed Therapy
Arm/Group | R-CHOP x 3 | R-CHOP x 6 | PET-negative: R-CHOP x 1 | PET-positive: IFRT + Yttrium-90 Ibritumomab Tiuxetan (Zevalin®)
Started | 0 | 0 | 137 | 12
Eligible and Evaluable | 0 | 0 | 113 | 12
Completed | 0 | 0 | 111 | 12
Not Completed | 0 | 0 | 26 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Refusal unrelated to adverse event | 0 | 0 | 1 | 0
Not completed — Ineligible | 0 | 0 | 24 | 0

BASELINE CHARACTERISTICS:
Population: Eligible and evaluable patients were included. The patient who was upstaged at baseline by PET/CT was not included.
Arm/Group | R-CHOP x 3
Number analyzed (Participants) | 132
Age, Continuous [Median (Full Range); unit: years] | 62 [18 to 86]
Age, Customized [Count of Participants; unit: Participants]
  Age > 60 years | 71
  Age <= 60 years | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 121
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 115
  More than one race | 0
  Unknown or Not Reported | 3
Zubrod Performance Status [Count of Participants; unit: Participants] — Grade 0: Fully active; able to carry on all pre-disease activities without restriction.
  Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  Grade 2: Ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  Grade 3: Capable of only limited self-care; confined to bed or chair more than 50% of waking hours.
  Grade 4: Completely disabled; cannot carry on any self-care; totally confined to bed or chair.
  Participants
    0 | 89
    1 | 39
    2 | 4
Stage [Count of Participants; unit: Participants] — Ann Arbor Classification (AJCC Manual for Staging of Cancer, 7th ed., 2010)
  Stage I: Involvement of a single lymph node region (I) or localized involvement of a single extralymphatic organ or site (IE).
  Stage II: Involvement of two or more lymph node regions on the same side of the diaphragm (II) or localized involvement of a single associated extralymphatic organ or site and its regional lymph nodes with or without other lymph node lesions on the same side of the diaphram (IIE).
  Participants
    Stage I | 82
    Stage II | 50
Symptoms [Count of Participants; unit: Participants] — A = Asymptomatic
  B = Fever, sweats, weight loss > 10% of body weight
  Participants
    A | 109
    B | 23
Elevated Lactate Dehydrogenase (LDH) [Count of Participants; unit: Participants]
  Yes | 19
  No | 113
Extranodal Involvement [Count of Participants; unit: Participants]
  Yes | 57
  No | 75
Stage-modified International Prognostic Index risk factors [Count of Participants; unit: Participants] — One point is assigned for each of the following statements that is true:
  1. Age (over 60)
  2. Performance status 2
  3. LDH greater than institutional upper limit of normal
  4. Stage II Disease
  Participants
    0 | 35
    1 | 55
    2 | 37
    3 | 5
Histologic Subtype [Count of Participants; unit: Participants]
  Diffuse large B-cell lymphoma, NOS | 95
  High-grade B-cell lymphoma with MYC and BCL2 or/and BCL6 rearrangements | 4
  High-grade B-cell lymphoma, NOS | 22
  T cell/histiocyte-rich large B-cell lymphoma | 2
  Central pathologic review not performed | 9
Cell of Origin by Lymph2Cx [Count of Participants; unit: Participants] — GCB: germinal center B-cell
  ABC: activated B-cell Population: Cell of origin by Lymph2Cx was assessable in 87 patients
  Participants
    number analyzed (Participants) | 87
    GCB | 59
    ABC | 20
    Unclassifiable | 8
Double protein expressors (DPE) [Count of Participants; unit: Participants] — Double protein expressor (DPE) status is defined as having both positive MYC staining of at least 40% and BCL2 staining of at least 50% of malignant cells on immunohistochemistry slides Population: Double protein expressor status was determined in 123 patients
  Participants
    number analyzed (Participants) | 123
    DPE | 21
    Non-DPE | 97
    Indeterminate | 5

OUTCOME MEASURES:

1. Primary Outcome: Five-year Progression-free Survival (PFS) Rate in Patients With Newly Diagnosed Limited Stage Diffuse Large B-cell Lymphoma (DLBCL)
Description: Measured from date of registration to date of first observation of progressive disease, or death due to any cause. Patients last known to be alive without report of progression or relapse are censored at date of last contact.
  Progressions is defined using the 2007 revised Cheson et. Al. criteria, as ≥50% increase in the sum of the products of diameters (SPD) of target measurable lesions, appearance of any new bone marrow involvement, or appearance of any new lesion >1.5 cm in the longest axis.
Time Frame: up to 5 years
Population: Eligible and evaluable patients were included in the analysis. The patient who was upstaged at baseline by PET/CT was not included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- R-CHOP x 3 Followed by PET-directed Therapy: R-CHOP x 3: Chemotherapy for up to 3 cycles, 21 days/per cycle, with R-CHOP
  For each cycle, R-CHOP therapy included:
  Rituximab: 375 mg/m^2 IV administration on Day 1
  Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  Doxorubicin: 50 mg/m^2 IV administration on Day 1
  Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  Prednisone: 100 mg administered orally on Days 1 through 5
  PET-directed therapy included:
  PET-negative: R-CHOP x 1 PET-positive: IFRT + Yttrium-90 ibritumomab tiuxetan
  R-CHOP x 1: 1 cycle of R-CHOP, 21 days/cycle
  Rituximab: 375 mg/m^2 IV administration on Day 1
  Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  Doxorubicin: 50 mg/m^2 IV administration on Day 1
  Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  Prednisone: 100 mg administered orally on Days 1 through 5
  IFRT + Yttrium-90 ibritumomab tiuxetan included:
  IFRT: 180 cGy/day for a minimum dose of 3600 cGy and a maximum of dose of 4500 cGy
  Rituximab: 250 mg/m^2 IV administration on Day 1 then 7, 8, or 9
  Yttrium-90 ibritumomab tiuxetan: 0.4 mCi/kg or 0.3 mCi/kg, absolute maximum allowable dose of 32.0 mCi, 10 min IV infusion, on Day 7, 8 or 9
Arm/Group | R-CHOP x 3 Followed by PET-directed Therapy
Number analyzed (Participants) | 132
percentage of participants | 87 [79 to 92]

2. Secondary Outcome: Progression-free Survival (PFS) Within the PET+ and PET- Subgroups of Patients With Newly Diagnosed Limited-stage Diffuse Large B-Cell Lymphoma (DLBCL)
Description: Measured from date of interim positron emission tomography (PET)/computed tomography scan to date of first observation of progressive disease, or death due to any cause. Patients last known to be alive without report of progression or relapse are censored at date of last contact.
Time Frame: up to 5 years
Population: Eligible and evaluable patients who had interim PET/CT performed were included in the analysis. The patient who was upstaged at baseline by PET/CT was not included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Interim PET-negative: Interim PET/CT scan was performed on Day 15-18 of Cycle 3 of R-CHOP chemotherapy. PET/CT scans were centrally reviewed and scored.
  Negative:
  1. no uptake
  2. uptake ≤ mediastinum
  3. uptake > mediastinum but ≤ liver
- Interim PET-positive: Interim PET/CT scan was performed on Day 15-18 of Cycle 3 of R-CHOP chemotherapy. PET/CT scans were centrally reviewed and scored.
  Positive:
  4 uptake > liver in some sites even if uptake ≤ liver or mediastinum at other sites 5 uptake > liver in over 90% of sites or development of new uptake consistent with progressive disease
Arm/Group | Interim PET-negative | Interim PET-positive
Number analyzed (Participants) | 114 | 14
percentage of participants | 89 [80 to 94] | 86 [54 to 96]

3. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: up to 4 months or time of disease progression.
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 4.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Groups:
- PET-positive: IFRT + Yttrium-90 Ibritumomab Tiuxetan (Zevalin®: Patients start Involved-Field Radiation Therapy (IFRT) as soon as possible after the Day 15-18 PET/CT scan that follows Cycle 3 of R-CHOP, but no later than Day 35 after initiation of Cycle 3 of R-CHOP. Zevalin® treatment begins 3-6 weeks after Radiation Therapy is completed.
  Radiation Therapy included:
  IFRT:180 cGy/day for a minimum dose of 3600 cGy and a maximum of dose of 4500 cGy
  Radioimmunotherapy included:
  Rituximab: 250 mg/m^2 IV administration on Day 1 then 7, 8, or 9
  Yttrium-90 ibritumomab tiuxetan: 0.4 mCi/kg or 0.3 mCi/kg, absolute maximum allowable dose of 32.0 mCi, 10 min IV infusion, on Day 7, 8 or 9
Arm/Group | R-CHOP x 3 | R-CHOP x 6 | PET-negative: R-CHOP x 1 | PET-positive: IFRT + Yttrium-90 Ibritumomab Tiuxetan (Zevalin®
Number analyzed (Participants) | 132 | 1 | 113 | 12
Participants
  Alanine aminotransferase increased | 0 | 0 | 1 | 0
  Anemia | 7 | 0 | 2 | 1
  Anorexia | 1 | 0 | 1 | 0
  Bone pain | 1 | 0 | 0 | 0
  CD4 lymphocytes decreased | 1 | 0 | 0 | 0
  Catheter related infection | 1 | 0 | 0 | 0
  Cough | 1 | 0 | 0 | 0
  Diarrhea | 2 | 0 | 0 | 0
  Dyspnea | 3 | 0 | 0 | 0
  Edema limbs | 1 | 0 | 0 | 0
  Endocrine disorders - Other, specify | 1 | 0 | 0 | 0
  Fall | 0 | 0 | 1 | 0
  Fatigue | 3 | 0 | 1 | 0
  Febrile neutropenia | 13 | 0 | 2 | 0
  Generalized muscle weakness | 1 | 0 | 0 | 0
  Hyperglycemia | 3 | 0 | 1 | 0
  Hypertension | 1 | 0 | 0 | 0
  Hypocalcemia | 0 | 0 | 1 | 0
  Hypokalemia | 2 | 0 | 1 | 0
  Hyponatremia | 1 | 0 | 1 | 0
  Hypotension | 0 | 0 | 1 | 0
  Hypoxia | 0 | 0 | 2 | 0
  Leukemia secondary to oncology chemotherapy | 0 | 0 | 1 | 0
  Lung infection | 2 | 0 | 0 | 0
  Lymphocyte count decreased | 16 | 0 | 9 | 2
  Nausea | 1 | 0 | 0 | 0
  Nervous system disorders - Other, specify | 0 | 0 | 1 | 0
  Neutrophil count decreased | 34 | 0 | 11 | 2
  Peripheral sensory neuropathy | 1 | 0 | 1 | 0
  Platelet count decreased | 5 | 0 | 4 | 3
  Resp, thoracic and mediastinal disorders - Other | 0 | 0 | 1 | 0
  Sepsis | 2 | 0 | 0 | 0
  Skin infection | 1 | 0 | 1 | 0
  Stroke | 1 | 0 | 0 | 0
  Thromboembolic event | 0 | 0 | 1 | 0
  Urinary tract infection | 3 | 0 | 0 | 0
  Weight loss | 0 | 0 | 1 | 0
  White blood cell decreased | 26 | 0 | 12 | 2

4. Secondary Outcome: Overall Survival of Patients With Newly Diagnosed Limited-stage Diffuse Large B-Cell Lymphoma (DLBCL)
Description: Measured from date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: up to 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | R-CHOP x 3 Followed by PET-directed Therapy
Number analyzed (Participants) | 132
percentage of participants | 89 [82 to 93]

5. Secondary Outcome: Response Rates in Patients With Newly Diagnosed Limited Stage Diffuse Large B-cell Lymphoma Using PET/CT Scan to Direct Therapy After 3 Cycles of R-CHOP
Description: Complete Response (CR) is a complete disappearance of all disease with the exception of the following. If no PET scan or when the PET scan was positive before therapy, a post-treatment residual mass of any size is permitted if it is PET negative. If the PET scan was negative before therapy, all nodal masses at baseline must have regressed. No new lesions. Previously enlarged organs must have regressed and not be palpable. Bone marrow (BM) must be negative if positive at baseline. Normalization of markers. Partial Response (PR) is a 50% decrease in the sum of products of greatest diameters (SPD) for up to 6 identified dominant lesions, including spleenic and hepatic nodules from baseline. No new lesions and no increase in the size of liver, spleen or other nodes. If PET scan or when the PET scan was positive before therapy, PET should be positive in at least one previously involved site.
Time Frame: Up to 4 months
Population: Eligible and evaluable patients who treated with PET-directed therapy based on FDG-PET imaging after 3 cycles of R-CHOP were included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- R-CHOP x 3 Followed by R-CHOP x 1 in Interim PET-negative Patients: R-CHOP x 3: Chemotherapy for up to 3 cycles, 21 days/per cycle, with R-CHOP
  For each cycle, R-CHOP therapy included:
  Rituximab: 375 mg/m^2 IV administration on Day 1
  Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  Doxorubicin: 50 mg/m^2 IV administration on Day 1
  Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  Prednisone: 100 mg administered orally on Days 1 through 5
  PET-directed therapy included:
  PET-negative: R-CHOP x 1
  R-CHOP x 1: 1 cycle of R-CHOP, 21 days/cycle
  Rituximab: 375 mg/m^2 IV administration on Day 1
  Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  Doxorubicin: 50 mg/m^2 IV administration on Day 1
  Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  Prednisone: 100 mg administered orally on Days 1 through 5
- R-CHOP x 3 Followed by IFRT + Yttrium-90 Ibritumomab Tiuxetan in Interim PET-positive Patients: R-CHOP x 3: Chemotherapy for up to 3 cycles, 21 days/per cycle, with R-CHOP
  For each cycle, R-CHOP therapy included:
  Rituximab: 375 mg/m^2 IV administration on Day 1
  Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  Doxorubicin: 50 mg/m^2 IV administration on Day 1
  Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  Prednisone: 100 mg administered orally on Days 1 through 5
  PET-directed therapy included:
  PET-positive: IFRT + Yttrium-90 ibritumomab tiuxetan
  IFRT: 180 cGy/day for a minimum dose of 3600 cGy and a maximum of dose of 4500 cGy
  Rituximab: 250 mg/m^2 IV administration on Day 1 then 7, 8, or 9
  Yttrium-90 ibritumomab tiuxetan: 0.4 mCi/kg or 0.3 mCi/kg, absolute maximum allowable dose of 32.0 mCi, 10 min IV infusion, on Day 7, 8 or 9
Arm/Group | R-CHOP x 3 Followed by R-CHOP x 1 in Interim PET-negative Patients | R-CHOP x 3 Followed by IFRT + Yttrium-90 Ibritumomab Tiuxetan in Interim PET-positive Patients
Number analyzed (Participants) | 113 | 12
Participants
  Complete Response | 112 | 8
  Partial Response | 0 | 4
  Inadequate Assessment | 1 | 0

6. Secondary Outcome: Association of Germinal Center B-cell Subtype (GCB) vs Stromal-1 vs Stromal-2 Gene Expression Signatures With PFS or Overall Survival.
Description: Formalin-fixed, paraffin-embedded tissue from the diagnostic biopsy is collected and used to determine germinal center B-cell (GCB) phenotype. GCB subtype of DLBCL is defined by gene-expression profiling that is performed using quantitative nuclease protection assay (qNPA).
  Data for this outcome measure is not available at this time. We expect this data to be available by December 2025.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: up to 4 months or time of disease progression
Description: The total number or participants at risk in this section is the number or participants in each arm that are eligible and evaluable.
Groups:
- PET-negative: R-CHOP x 1: Chemotherapy for 1 cycle, 21 days/per cycle, with R-CHOP
  R-CHOP therapy included:
  Rituximab: 375 mg/m^2 IV administration on Day 1
  Cyclophosphamide: 750 mg/m^2 IV administration on Day 1
  Doxorubicin: 50 mg/m^2 IV administration on Day 1
  Vincristine: 1.4 mg/m^2 (maximum 2 mg) IV administration on Day 1
  Prednisone: 100 mg administered orally on Days 1 through 5 2
Arm/Group | R-CHOP x 3 | R-CHOP x 6 | PET-negative: R-CHOP x 1 | PET-positive: IFRT + Yttrium-90 Ibritumomab Tiuxetan (Zevalin®)
All-Cause Mortality (participants affected / at risk) | 1/132 | 0/1 | 1/113 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/132 | 0/1 | 2/113 | 0/12
Other Adverse Events (participants affected / at risk) | 130/132 | 1/1 | 105/113 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R-CHOP x 3 (N=132) | R-CHOP x 6 (N=1) | PET-negative: R-CHOP x 1 (N=113) | PET-positive: IFRT + Yttrium-90 Ibritumomab Tiuxetan (Zevalin®) (N=12)
Sudden death NOS (General disorders) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R-CHOP x 3 (N=132) | R-CHOP x 6 (N=1) | PET-negative: R-CHOP x 1 (N=113) | PET-positive: IFRT + Yttrium-90 Ibritumomab Tiuxetan (Zevalin®) (N=12)
Anemia (Blood and lymphatic system disorders) | 68 | 1 | 45 | 5
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 13 | 0 | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 5 | 0 | 3 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Endocrine disorders-Other (Endocrine disorders) | 1 | 0 | 0 | 0
Blurred vision (Eye disorders) | 5 | 0 | 2 | 1
Eye disorders-Other (Eye disorders) | 1 | 0 | 2 | 0
Eye pain (Eye disorders) | 1 | 0 | 1 | 0
Floaters (Eye disorders) | 1 | 0 | 1 | 0
Watering eyes (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 0 | 2 | 2
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Bloating (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 52 | 1 | 7 | 1
Diarrhea (Gastrointestinal disorders) | 19 | 0 | 7 | 2
Dry mouth (Gastrointestinal disorders) | 12 | 0 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 15 | 0 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 4 | 0 | 1 | 4
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 | 0 | 5 | 0
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 19 | 1 | 4 | 1
Nausea (Gastrointestinal disorders) | 60 | 1 | 11 | 2
Oral pain (Gastrointestinal disorders) | 4 | 0 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 13 | 1 | 2 | 0
Chills (General disorders) | 9 | 0 | 2 | 1
Edema face (General disorders) | 2 | 0 | 0 | 0
Edema limbs (General disorders) | 11 | 1 | 4 | 0
Facial pain (General disorders) | 3 | 0 | 0 | 0
Fatigue (General disorders) | 90 | 1 | 51 | 7
Fever (General disorders) | 12 | 0 | 2 | 0
Flu like symptoms (General disorders) | 3 | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
General disorders and admin site conditions - Other (General disorders) | 3 | 0 | 1 | 0
Infusion related reaction (General disorders) | 12 | 0 | 0 | 0
Injection site reaction (General disorders) | 2 | 0 | 0 | 0
Localized edema (General disorders) | 3 | 0 | 2 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 3 | 0 | 1 | 0
Pain (General disorders) | 4 | 0 | 7 | 0
Allergic reaction (Immune system disorders) | 5 | 0 | 0 | 0
Autoimmune disorder (Immune system disorders) | 1 | 0 | 0 | 0
Bronchial infection (Infections and infestations) | 1 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 1 | 0
Eye infection (Infections and infestations) | 2 | 0 | 0 | 0
Gum infection (Infections and infestations) | 1 | 0 | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0 | 1 | 0
Infections and infestations-Other (Infections and infestations) | 0 | 0 | 3 | 0
Lip infection (Infections and infestations) | 2 | 0 | 0 | 0
Lung infection (Infections and infestations) | 2 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 1 | 0
Papulopustular rash (Infections and infestations) | 1 | 0 | 0 | 0
Peripheral nerve infection (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0
Skin infection (Infections and infestations) | 6 | 0 | 6 | 0
Upper respiratory infection (Infections and infestations) | 9 | 0 | 5 | 1
Urinary tract infection (Infections and infestations) | 10 | 0 | 1 | 1
Vaginal infection (Infections and infestations) | 2 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 26 | 0 | 16 | 1
Alkaline phosphatase increased (Investigations) | 5 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 15 | 0 | 9 | 1
Blood bilirubin increased (Investigations) | 3 | 0 | 1 | 0
CD4 lymphocytes decreased (Investigations) | 2 | 0 | 0 | 0
Carbon monoxide diffusing capacity decreased (Investigations) | 1 | 0 | 0 | 0
Cardiac troponin I increased (Investigations) | 1 | 0 | 0 | 0
Cholesterol high (Investigations) | 1 | 0 | 0 | 0
Creatinine increased (Investigations) | 7 | 0 | 4 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0
Fibrinogen decreased (Investigations) | 1 | 0 | 0 | 0
Forced expiratory volume decreased (Investigations) | 1 | 0 | 0 | 0
Hemoglobin increased (Investigations) | 1 | 0 | 0 | 0
INR increased (Investigations) | 3 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 57 | 1 | 44 | 4
Neutrophil count decreased (Investigations) | 46 | 0 | 16 | 5
Platelet count decreased (Investigations) | 23 | 1 | 18 | 4
Vital capacity abnormal (Investigations) | 1 | 0 | 0 | 0
Weight gain (Investigations) | 2 | 1 | 3 | 0
Weight loss (Investigations) | 5 | 0 | 4 | 3
White blood cell decreased (Investigations) | 49 | 1 | 34 | 5
Anorexia (Metabolism and nutrition disorders) | 13 | 1 | 5 | 4
Dehydration (Metabolism and nutrition disorders) | 8 | 0 | 1 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 24 | 0 | 12 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypernatremia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 19 | 1 | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 11 | 0 | 4 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 11 | 0 | 5 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 10 | 0 | 5 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 0 | 10 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 0 | 4 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 21 | 1 | 2 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 1 | 4 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 1 | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 7 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 1 | 0
Concentration impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 11 | 0 | 2 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 15 | 0 | 8 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 17 | 1 | 2 | 0
Memory impairment (Nervous system disorders) | 2 | 0 | 1 | 0
Movements involuntary (Nervous system disorders) | 1 | 0 | 0 | 0
Nervous system disorders-Other (Nervous system disorders) | 1 | 0 | 1 | 1
Paresthesia (Nervous system disorders) | 4 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 5 | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 35 | 0 | 21 | 2
Presyncope (Nervous system disorders) | 2 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 2 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 12 | 1 | 1 | 1
Confusion (Psychiatric disorders) | 4 | 0 | 2 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 3 | 1 | 0 | 1
Hallucinations (Psychiatric disorders) | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 22 | 0 | 3 | 2
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 2 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal and urinary disorders-Other (Renal and urinary disorders) | 2 | 0 | 1 | 0
Renal calculi (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 12 | 0 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 3 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 3 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 1 | 0
Urinary urgency (Renal and urinary disorders) | 2 | 0 | 0 | 0
Urine discoloration (Renal and urinary disorders) | 1 | 0 | 1 | 0
Irregular menstruation (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 1 | 10 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 | 1 | 7 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1 | 0
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 2 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 53 | 1 | 21 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 1 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 3 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 1 | 1 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 9 | 0 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hot flashes (Vascular disorders) | 4 | 0 | 4 | 0
Hypertension (Vascular disorders) | 19 | 1 | 11 | 0
Hypotension (Vascular disorders) | 4 | 0 | 1 | 0
Lymphedema (Vascular disorders) | 1 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 1 | 0
Superficial thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 2 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT01359592/Prot_SAP_ICF_000.pdf